CLINICAL TRIAL: NCT05067179
Title: Analysis of Human ALS Tissues and Registry of ALS Patients
Status: Recruiting | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Principal Investigator, Jeffrey A Loeb, Neurology and Rehabilitation Department Chair, University of Illinois at Chicago
Other Study IDs: 2013-0748
Record Dates: First submitted 2021-09-07; First posted 2021-10-05 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis (ALS); Lou Gehrig's Disease; Neurodegenerative Diseases; Neuromuscular Diseases; Nervous System Diseases
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases; Neuromuscular Diseases; Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tissue from different body regions including brain, spinal cord, nerve and muscle.
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS), often referred to as Lou Gehrig's Disease, is a progressive, terminal condition of muscle weakness that is associated with degeneration of neurons in the spinal cord and brain. This devastating disorder afflicts people in the prime of their lives. At the present time, there are no cures for this disorder, and current treatments are marginal at best. Despite years of intensive research, a fundamental understanding of this disease is still lacking. There is a need to identify both reliable markers of disease progression and effective treatments. The goal of this research is to bring a greater understanding of ALS patients closer to the research studies that can lead to new hypotheses and approaches.

DETAILED DESCRIPTION:
Patients will be approached during in-person or phone/online appointments and asked their consent to enter information and results from their physical examinations, electrodiagnostic testing, and other testing done as a standard of care and into a database to monitor disease progression and use them for research purposes. Also, the patients will be asked for consent to undergo a MRI scan.

In a second informed consent form, patients will be enrolled to perform a rapid postmortem autopsy and have the tissue banked for research purposes. It is important to keep the consents separate because some patients may not consent to this postmortem study, but would consent to the premortem studies.

The information gained from the premortem studies will be used during the postmortem examination to select tissue for further processing. Tissue from different regions, including brain, spinal cord, nerve and muscle will be processed in parallel for cellular and molecular analyses that include histology, immunostaining, in situ hybridization, protein, RNA, and small molecule analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Established diagnosis of ALS
* Able and willing to give written informed consent and must authorize release and use of protected health information

Exclusion Criteria:

* Patients below the age of 18
* No diagnosis of ALS

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged > 18 years with a diagnosis of ALS being seen at the Neuromuscular Center Clinics, University of Illinois at Chicago
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Imaging biomarkers | Within 6 months of participant enrollment
  High resolution 3T MRI T1, T2/FLAIR, DWI, SWI, MRS, and MT sequences at the cervical, thoracic, and lumbar spine and brainstem will be used to identify individual and combinatorial (of each sequence) changes to be used as clinical biomarkers of progression in cases with focal disease onset and spread. These will be compared to histologic and genomic changes in rapid postmortem tissues in the same areas. High resolution T1-weighted imaging is preferred for anatomical structure morphometry. The hypothesis is that spinal cord cross-sectional area decreases over time may be a sensitive MRI parameter to detect progression and respiratory distress. The aim is to develop a highly sensitive and specific, non-invasive measure of ALS progression in the spinal cord using a multi-parametric measurement scheme. Image sequences will be attained and a combinatorial statistical analysis performed to find the best biomarker of progression that could differ regardless of upper motor neuron involvement.
Molecular biomarkers | Within 12 months of participant's passing
  Tissue analyses will be performed to identify differentially expressed genes and histological differences from a rapid postmortem analysis of human ALS tissues from the same spinal cord levels and brainstem imaged on MRI, using an initial genomic analysis (RNAseq). Clinically meaningful biomarkers for disease progression will be validated through bioinformatics and confirmatory studies on human tissues and linked to imaging and clinical findings. Further analysis will look for differences in those with and without upper motor neuron involvement and for those taking or not taking drugs. Tissues will be stored for future studies.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Loeb, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States